CLINICAL TRIAL: NCT06340503
Title: Evaluating a Physical Activity Index for Assessment and Counseling for Breast and Colon Cancer Survivors in Clinical Practice
Brief Title: Evaluating a Physical Activity Index for Assessment and Counseling for Breast and Colon Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00111331; WFBCCC 01123 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Physical activity; Exercise coaching
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Motor Activity | interventions — Interviews as Topic; Health Surveys

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants randomized into the exercise group will receive a pre-exercise screening call about two weeks after enrolling into the study and complete the six (6) study visits and pre-determined test and procedures for the patient intervention arm.
  Interventions: Device: Research-grade accelerometer; Other: National Comprehensive Cancer Network (NCCN) Education Materials; Device: Garmin Vivofit activity tracker; Other: Exercise Consultation Calls; Other: Interview; Other: Physical Activity Index Assessment (Intervention Arm); Other: Health Surveys
- Delayed Exercise Group (Active Comparator): Participants randomized to the delayed exercise group, will have vitals collected and complete surveys at the first (baseline), 3-month, and 6-month visits pre-determined test and procedures for the waitlist control arm. The pre-exercise consultation will begin after the 6-month visit.
  Interventions: Device: Research-grade accelerometer; Other: National Comprehensive Cancer Network (NCCN) Education Materials; Device: Garmin Vivofit activity tracker; Other: Interview; Other: Physical Activity Index Assessment (Control Arm); Other: Health Surveys

INTERVENTIONS:
Device: Research-grade accelerometer — Participants will be instructed to wear device for 7 days prior to each visit and to bring the device to each visit. Study staff will extract data from the device within 14 days after each appointment and return the device to patients by mail.
Other: National Comprehensive Cancer Network (NCCN) Education Materials — The NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®) are comprised of recommendations for the prevention, diagnosis, and management of malignancies across the continuum of care.
Device: Garmin Vivofit activity tracker — This device can automatically capture and classify different physical activities such as walking, running, biking, swimming and using an elliptical.
Other: Exercise Consultation Calls — The intervention group will receive five monthly exercise consultation calls with an exercise coach in between clinical visits and be provided with an exercise log for their personal use
  Arms: Exercise Group
Other: Interview — The interviews will be conducted by a trained Q-PRO interviewer and audio recorded. Interviews are expected to last approximately 30 minutes. Discussion will include acceptability of the PAI intervention, related tools, and clinical experiences and will help shape/inform refinements need for a larger efficacy trial
Other: Physical Activity Index Assessment (Intervention Arm) — Assessment will capture frequency and time spent in strenuous, moderate, and mild PA over the past 7 days. Survivors also report hours of TV or similar sedentary screen time per week as a measure of sedentary behavior. Completed at months 1, 3, 6, 9 and 12 while on study
  Arms: Exercise Group
Other: Physical Activity Index Assessment (Control Arm) — Assessment will capture frequency and time spent in strenuous, moderate, and mild PA over the past 7 days. Survivors also report hours of TV or similar sedentary screen time per week as a measure of sedentary behavior. Completed at months 6, 9 and 12 while on study.
  Arms: Delayed Exercise Group
Other: Health Surveys — Various health surveys will be completed to assess participant health and physical activities.

SUMMARY:
The purpose of this research study is to determine whether using the physical activity index screener, exercise coaching, and self-monitoring will increase physical activity and reduce time spent sitting or being inactive in patients who had breast or colon cancer.

DETAILED DESCRIPTION:
To assess the feasibility (participation rate, adherence, and retention) of the Physical Activity Index (PAI) intervention in breast and colon cancer survivors supported by exercise coaching and self-monitoring tools.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of breast or colon cancer (stages 0-III) diagnosed within the last three years prior to enrollment.
* Completed primary treatment (surgery, chemotherapy, and/or radiation) at least 3 months prior to enrollment.
* At least 50 years of age or older.
* Access to internet or cellular plan for video calls.
* Being willing and able to comply with the approved protocol and able to sign an IRB-approved informed consent document directly, remotely or via electronic consent.
* Able to read and speak English

Exclusion Criteria:

* Participants with metastatic disease.
* Participants with recurrence or diagnosis of a different cancer.
* Participants receiving treatment other than maintenance therapy for their primary cancer (breast or colon).
* Participants has prior conditions that contraindicate exercise as determined by treating physician.
* Participants has gross cognitive impairment as determined by treating physician.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Eligible Participants - Participation Rate | 17 months
  Participation will be measured by the number of eligible participants who agree to participate. Investigators will calculate 95% confidence interval for each of the feasibility measures to determine the range of estimates that are consistent with the data.
Percentage of Participants to Complete Exercise Sessions - Adherence | 17 months
  Adherence will be measured by the percent of participants who complete at least 3 out 5 exercise sessions. Investigators will calculate 95% confidence interval for each of the feasibility measures to determine the range of estimates that are consistent with the data.
Number of Participants Who Complete Study Questionnaires - Retention | At baseline and up to 17 months
  Retention will be defined as the number of participants who complete study questionnaires at baseline and one follow-up timepoint. Investigators will calculate 95% confidence interval for each of the feasibility measures to determine the range of estimates that are consistent with the data.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Bluethmann, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No